CLINICAL TRIAL: NCT01156428
Title: Transcriptional Profiling of Kidney Tissue Obtained From Patients With Newly Identified Proteinuria, Nephrotic Syndrome or Nephritic Syndrome
Brief Title: Inflammatory and Immune Profiling of Kidney Tissue Obtained From Patients With Newly Diagnosed Kidney Disease
Status: Completed | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0908010598
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Proteinuria; Kidney Injury; Chronic Kidney Disease
Keywords: Nephritic syndrome; Nephrotic syndrome; Proteinuria; Acute kidney injury; Chronic kidney disease; Lupus nephritis
MeSH Terms: conditions — Proteinuria; Renal Insufficiency, Chronic; Nephrotic Syndrome; Acute Kidney Injury; Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, urine, kidney tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Subjects (normal volunteers): Control kidney specimens will be obtained from donor transplant kidneys or nephrectomy specimens performed on patients undergoing nephrectomy for the clinical indication of an identified renal mass.
  In the case of donor transplant kidneys, the renal biopsy will be conducted during the act of living donor nephrectomy and transplantation.
  In the case of renal mass nephrectomies, representative "normal" tissue will be obtained from the nephrectomized kidney at a site distant from the renal mass.
- Renal Disease Subjects: Patients who require a renal biopsy based upon clinical indications such as proteinuria, hematuria, acute renal failure (ARF) of unclear etiology, chronic kidney disease of unclear etiology, nephrotic syndrome, nephritic syndrome, suspected lupus nephritis or any other medically warranted indication for a biopsy.

SUMMARY:
This study will evaluate in patients with kidney disease, the role that certain inflammatory and immune mediators play in promoting kidney damage. The investigators hypothesize that certain mediators, (identified in the serum, urine and renal biopsy tissue), of patients with a variety of different renal disease states will provide information regarding their clinical course and that inflammatory and immune patterns in the serum and urine of patients with kidney disease may yield predictive diagnostic information in place of a renal biopsy. The ability to detect and quantify these mediators may lead to earlier detection and treatment of kidney disease in order to prevent kidney failure and the requirement for renal replacement.

The study will evaluate serum, blood and urine collected over a one year period post kidney biopsy for the presence of inflammatory or immune mediators, which will be correlated with kidney pathology findings (gene signatures). These gene signatures will be compared to "normal" control specimens obtained from donor transplant kidneys or from normal kidney tissue obtained from patients who require their entire kidney removed for a tumor.

DETAILED DESCRIPTION:
The aim of the study is to evaluate in humans inflammatory and immune mediators that may play a role in kidney damage. The investigators hypothesize that certain inflammatory and immune mediators identified in the serum and/or urine of patients with a variety of different renal disease states will provide prognostic information regarding their clinical course. Furthermore, we hypothesize that RNA transcriptional profiling of renal biopsy specimens will identify gene array patterns that provide prognostic information for various disease states. Lastly, we hypothesize that patterns of inflammatory and immune mediators identified in serum and/or urine may yield predictive diagnostic information in lieu of renal biopsy. The ability to detect and quantify these mediators may lead to earlier detection and treatment prior to the progression of Chronic Kidney Disease (CKD) to stage 4 and/or 5.

The study will evaluate serially collected serum, blood and urine over a one-year period post kidney biopsy for both the presence of inflammatory or immune mediators. The blood, serum and urine inflammatory and immune mediators will be correlated with the kidney pathology gene signature. Note that all of the biopsies are conducted based upon clinical indication and not for the purpose of the study.

Renal pathology gene signatures obtained from study subjects will be compared to "normal" control specimens. Normal specimens will be obtained from donor transplant kidneys or nephrectomy specimens performed on patients undergoing nephrectomy for the clinical indication of an identified renal mass. Representative "normal" tissue will be obtained from the nephrectomized kidney at a site distant from the renal mass.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18 years to 90 years old
* Any subject with pre-existing clinical indication of a kidney biopsy including, but not limited to, nephritic syndrome, nephritic syndrome or proteinuric disease state. Additionally, kidney transplant donors will be included for purpose of obtaining control tissue.
* Willing and able to give consent
* Additionally, kidney transplant donors and patients requiring nephrectomy for removal of renal mass will be included for purpose of obtaining control tissue.

Exclusion Criteria:

* Subjects on longstanding immunosuppressive agents (empiric initiation of glucocorticoid therapy within 48 hours prior to kidney biopsy is acceptable)
* Kidney transplant recipient
* Inability to follow-up for future protocol laboratory evaluation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject with pre-existing clinical indication for a kidney biopsy including, but not limited to, nephritic syndrome, nephritic syndrome or proteinuric disease state.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2010-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The deviation from the norm of whole blood, serum and urine inflammatory and immune mediators, renal biopsy gene signature patterns in subjects with a variety of biopsy proven renal conditions compared to normal subjects. | 12 months
  To determine the deviation from the norm of blood and urine inflammatory and immune mediators in subjects that have undergone renal biopsy for clinical indication with resultant biopsy diagnosed renal conditions.
  To determine the correlation of serum, whole blood and urine inflammatory and immune mediators with the renal pathologic diagnosis as well as the gene signature of the given pathology.

SECONDARY OUTCOMES:
Change over time of serum, whole blood and urine inflammatory and immune mediators. | 5 years
  Subjects clinical course and outcome will be followed over five years and related to change over time of serum, whole blood and urine inflammatory and immune mediators. This follow-up analysis may yield markers that correlate with therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Perlman, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States